CLINICAL TRIAL: NCT06794268
Title: Non-interventional Cohort Study of Patients Treated With Liso-cel (Lisocabtagene Maraleucel) for Relapsed/Refractory Follicular Lymphoma in the Postmarketing Setting
Brief Title: A Study to Patients With Relapsed/Refractory Follicular Lymphoma Treated With Liso-cel (Lisocabtagene Maraleucel) in the Post Marketing Setting
Status: Recruiting | Type: Observational
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CA082-1175
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving lisocabtagene maraleucel treatment
  Interventions: Biological: Lisocabtagene maraleucel

INTERVENTIONS:
Biological: Lisocabtagene maraleucel — As per product label

SUMMARY:
The purpose of this study is to characterise the long-term safety of lisocabtagene maraleucel, focusing on patients treated in the approved follicular lymphoma (FL) indication, and will be part of post-marketing liso-cel pharmacovigilance activities

ELIGIBILITY:
Inclusion Criteria:

• Participants must have been treated in the post-marketing setting with at least 1 infusion of lisocabtagene maraleucel (liso-cel) used for the treatment of relapsed/refractory (R/R) follicular lymphoma (FL), including FL Grade 1, Grade 2 and Grade 3a, within the FDA-approved indication and dosage per the United States Prescribing Information (USPI) and product specifications approved for commercial release in the USA

Exclusion Criteria:

* Participants known to be participating in investigational studies at the time of liso-cel, infusion
* Participants treated with liso-cel for the treatment of R/R FL Grade 3b
* Participants treated with non-conforming chimeric antigen receptor (CAR) T-cell product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adults with relapsed/refractory follicular lymphoma that are being treated with lisocabtagene maraleucel and are registered within the Center for International Blood and Marrow Transplant Research (CIBMTR) registry.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2044-08-31 (Estimated); Study Completion 2044-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) of interest | Up to 15 years
  AEs of interest include:
  * Secondary malignancies
  * Cytokine release syndrome (CRS) Grade ≥ 3
  * Neurotoxicity Grade ≥ 3
  * Prolonged cytopenias
  * Pregnancy outcome
  * Tumor lysis syndrome (TLS) Grade ≥ 3
  * Serious infections (ie, those requiring treatment)
  * Organ toxicities Grade ≥ 3
  * Hemophagocytic lymphohistiocytosis (HLH)/ macrophage activation syndrome (MAS)-like toxicities
  * Aggravated graft-versus-host disease (GvHD)
Incidence of other adverse events (AEs) of interest | Up to 15 years
  Other clinically important events that have not yet been identified as part of the liso-cel safety profile

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 15 years
Overall response rate (ORR) | Up to 15 years
Complete remission rate (CRR) | Up to 15 years
Duration of response (DOR) | Up to 15 years
Progression-free survival (PFS) | Up to 15 years
Time to next treatment (TTNT) | Up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- CIBMTR, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts